CLINICAL TRIAL: NCT05574842
Title: Effect of Double Duty Interventions on Double Burden of Malnutrition, Dietary Diversity Score, and Frequency of Morbidity Among Secondary School Adolescents in Central Ethiopia: Cluster Randomized Controlled Trial
Brief Title: The Effect of Double Duty Interventions on Double Burden of Malnutrition Among School Adolescents in Ethiopia
Acronym: DBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debre Berhan University (Other)
Collaborators: Jimma University (Other)
Responsible Party: Principal Investigator, Lemma Getacher, Principal Investigator, Debre Berhan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12/345/15
Record Dates: First submitted 2022-09-30; First posted 2022-10-12 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Malnutrition; Degree, Moderate; Diet Habit; Undernutrition; Overnutrition; Underweight; Overweight
Keywords: Double burden of malnutrition; Double-duty interventions; malnutrition; nutrition interventions
MeSH Terms: conditions — Malnutrition; Lymphoma, Follicular; Feeding Behavior; Overnutrition; Thinness; Overweight | interventions — Nutrition Assessment; Counseling

STUDY DESIGN:
Intervention Model Description: A two-arm parallel cluster randomized control trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Due to the nature of the double-duty interventions, participant allocation concealment will not be possible. However, data collectors, participants, and nutrition behavior change communicators will be blinded from the study hypotheses. Besides, by using and labeling a non-identifiable unique number, the data entry clerk will be blinded until data analysis will be finalized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will be received the double duty intervention through nutrition behavior change communication approach using a Health Belief Model.
  Interventions: Behavioral: Double duty interventions using nutrition behavior change communication approach
- Control (No Intervention): The control arm will not be received the double duty intervention, rather they receive the standard intervention given by the government.

INTERVENTIONS:
Behavioral: Double duty interventions using nutrition behavior change communication approach — The packages of the double-duty interventions were modified and adapted from the 2017 WHO policy brief report and Hawkes et al., 2020. These interventions are optimized strong education and nutrition behavior change communication focused on promotion of healthy diets (adequate adolescent nutrition, dietary diversity), physical activity (doing moderate intensity physical exercise, avoiding sitting for log time), prevent undue harm from energy-dense foods (avoiding Junk processed foods, avoiding fizzy sweetened drinks, street fast foods, chips, salt, sugar, fats etc.), and regulations on marketing foods from the customer side (e.g., buying of packed foods frequently).
  Other Names: Nutrition education and counselling (NEC), nutrition behavior change communication (NBCC)
  Arms: Intervention

SUMMARY:
The goal of this cluster randomized controlled trial is to determine the effect of double duty interventions on double burden of malnutrition, dietary diversity score, and frequency of morbidity among secondary school adolescents in Debre Berhan City, Ethiopia. The main aim is to answer the following questions.

1. What is the effect of double duty interventions on double burden of malnutrition among secondary school adolescents?
2. What is the effect of double duty interventions on dietary diversity score among secondary school adolescents?
3. What is the effect of double duty interventions on among secondary school adolescents?

DETAILED DESCRIPTION:
Introduction Double Burden of Malnutrition (DBM) is the simultaneous coexistence of undernutrition along with overweight and obesity within the same individuals, households, and populations at the national and international levels across the life course. For example, when DBM exists at the individual level, it can be occurring in the form of obesity with deficiency of one or more vitamins and minerals, or overweight in an adult who was stunted during childhood. Similarly, at the household level, it may be manifest in the forms of an overweight or anemic woman with underweight adolescents or grandparent. When it exists at the population level, the prevalence of both undernutrition and overweight/obesity can occur in the same community, nation, or region.

Adolescence is a critical period in the life-course of individuals next to infancy due to highly increased growth and development. It is ranging from 10 to 19 years and is a transition period from childhood to adulthood according to WHO. It is a period in which developmental effects related to puberty and brain development lead to new sets of diets, and also a time when increased nutrient intake is required for their rapid growth.

Every person obtains the social, physical, emotional, cognitive, and economic resources that are the groundwork for later life healthiness and welfare during adolescence. These resources outline paths of adolescents into the succeeding generations. Therefore, strategies, interventions, and investments in adolescent health and wellbeing bring benefits today, for decades to come, and for the next generation.

Double-duty interventions (DDIs) are interventions that have the potential to simultaneously tackle the burden of both undernutrition and overnutrition or diet-related NCDs in a comprehensive manner. These interventions can be achieved in three ways. First, though not harming the existing interventions on malnutrition. Second, by retrofitting the existing nutrition interventions to address all sorts of malnutrition. Third, through the development of de novo integrated interventions (starting from the beginning, anew, or a new) aimed at the DBM. These actions reflecting the shared drivers and platforms of contrasting forms of malnutrition.

Double-duty interventions also have the potential to improve nutrition outcomes across the spectrum of malnutrition through integrated initiatives, policies, and programs. It is not a zero-sum game in addressing contrasted and confounded forms of malnutrition in the global population. According to WHO 2017 policy brief, double-duty actions include about ten packages. These packages are categorized as health services packages, social safety nets packages, educational settings packages, agriculture, food systems, and food environments packages.

These selected potential candidates for double-duty interventions from each setting can be summarized into four points. These interventions are optimized strong education and nutrition behavior change communication focused on promotion of healthy diets (adequate adolescent nutrition, dietary diversity), physical activity (doing proper physical exercise, avoiding sitting for log time), prevent undue harm from energy-dense foods (avoiding junk processed foods, avoiding fizzy sweetened drinks, street fast foods, chips, salt, sugar etc.), and regulations on marketing foods from the customer side (e.g., buying of packed foods frequently). For this project, the most important and selected packages will be applied.

The final outcomes expected from this study are:

* The proportion of secondary school adolescents with double burden of malnutrition who have received the selected double-duty interventions (DDIs).
* The proportion of secondary school adolescents with high dietary diversity score (greater than or equal to 5 food groups from ten food groups) who have received the selected double-duty interventions (DDIs).
* The proportion of secondary school adolescents with frequency of morbidity who have received the selected double-duty interventions (DDIs).

Research Hypothesis of the Study

After this study has conducted, the following proposed expected outcomes will be achieved.

* The double-duty interventions will be decreased the double burden of malnutrition in adolescents.
* The double-duty interventions will be increased dietary diversity score of adolescents.
* The double-duty interventions will decrease the frequency of morbidity of adolescents.

Methods and Materials of the Study

Study area, period, and setting

This study will be conducted in Debre Berhan Regiopolitan City, North Shoa Zone, Amhara Region, Central Ethiopia. Debre Berhan Regiopolitan city is located 130 km away from Addis Ababa (the capital city of Ethiopia) and 690 km from Bahir Dar (the capital city of the Amhara region). It was founded by Emperor Zara Yakoob, and it is the capital city of North Shoa Zone of Amhara region. The city has coordinated with 9°41'N 39°32'E latitude and longitude, respectively. It is found at, 2840 m above sea level, which makes it the highest city of this size in Africa.

Study Design

This study will be used a six-month two-arm parallel design community-based cluster randomized controlled trial using clusters (kebeles) as a unit of randomization in the city.

ELIGIBILITY:
Inclusion Criteria:

* The study will be targeted secondary school adolescents in the study area.
* Secondary school adolescents who have followed their teaching learning process in the selected secondary schools for at least six months and above in the city during the study period will be included.
* Moreover, adolescents who had no intention of leaving the secondary schools until the end of the study will be included in this study.

Exclusion Criteria:

* Secondary school adolescents who will not be able to respond to an interview and who have physical disability including deformity such as kyphosis, scoliosis, and limb deformity which prevents standing erect will be excluded. Because it is not appropriate for anthropometric measurement.
* Moreover, participants who had confirmed diseases such as diabetes mellitus, hypertension etc., will be excluded from this study to improve the precision of anthropometric measurements and dietary practice.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 742 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Proportions of Double Burden of Malnutrition | six months [25 weeks]
  The proportion of secondary school adolescents with double burden of malnutrition who have received the selected double-duty interventions (DDIs) using an interviewer administered questionnaire.

SECONDARY OUTCOMES:
Proportions of High Dietary Diversity Score (taking ≥ 5 food groups from 10 food groups) | six months [25 weeks]
  The proportion of secondary school adolescents with high dietary diversity score (greater than or equal to 5 food groups from ten food groups) who have received the selected double-duty interventions (DDIs) using an interviewer administered questionnaire.
Proportions of Frequency of Morbidity | six months [25 weeks]
  The proportion of secondary school adolescents with frequency of morbidity who have received the selected double-duty interventions (DDIs) using an interviewer administered questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Debre Berhan University, Addis Ababa, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Yet, I have no plan to share IPD to other researchers.

REFERENCES:
- [Background] Kulkarni VS, Kulkarni VS, Gaiha R. "Double Burden of Malnutrition": Reexamining the Coexistence of Undernutrition and Overweight Among Women in India. Int J Health Serv. 2017 Jan;47(1):108-133. doi: 10.1177/0020731416664666. Epub 2016 Sep 15. PMID 27638762
- [Background] Azzopardi PS, Hearps SJC, Francis KL, Kennedy EC, Mokdad AH, Kassebaum NJ, Lim S, Irvine CMS, Vos T, Brown AD, Dogra S, Kinner SA, Kaoma NS, Naguib M, Reavley NJ, Requejo J, Santelli JS, Sawyer SM, Skirbekk V, Temmerman M, Tewhaiti-Smith J, Ward JL, Viner RM, Patton GC. Progress in adolescent health and wellbeing: tracking 12 headline indicators for 195 countries and territories, 1990-2016. Lancet. 2019 Mar 16;393(10176):1101-1118. doi: 10.1016/S0140-6736(18)32427-9. Epub 2019 Mar 12. PMID 30876706
- [Background] WHO. Guideline: Implementing Effective Actions for Improving Adolescent Nutrition [Internet]. 2018. Available from: http://apps.who.int/iris/bitstream/handle/10665/260297/9789241513708-eng.pdf%0Ajsessionid=19D1CBFA434795BA1645CC009FFE99A4?sequence=1
- [Background] Das JK, Salam RA, Thornburg KL, Prentice AM, Campisi S, Lassi ZS, Koletzko B, Bhutta ZA. Nutrition in adolescents: physiology, metabolism, and nutritional needs. Ann N Y Acad Sci. 2017 Apr;1393(1):21-33. doi: 10.1111/nyas.13330. PMID 28436102
- [Background] Nicholson A, Fawzi W, Canavan C, Keshavjee S. Advancing Global Nutrition for Adolescent and Family Health : Innovations in Research and Training. Proceedings of the Harvard Medical School Center for Global Health Delivery-Dubai. 2018, Dubai, United Arab Emirates. 2018. p. 1-75.
- [Background] Patton GC, Sawyer SM, Santelli JS, Ross DA, Afifi R, Allen NB, Arora M, Azzopardi P, Baldwin W, Bonell C, Kakuma R, Kennedy E, Mahon J, McGovern T, Mokdad AH, Patel V, Petroni S, Reavley N, Taiwo K, Waldfogel J, Wickremarathne D, Barroso C, Bhutta Z, Fatusi AO, Mattoo A, Diers J, Fang J, Ferguson J, Ssewamala F, Viner RM. Our future: a Lancet commission on adolescent health and wellbeing. Lancet. 2016 Jun 11;387(10036):2423-78. doi: 10.1016/S0140-6736(16)00579-1. Epub 2016 May 9. No abstract available. PMID 27174304
- [Background] Hargreaves D, Mates E, Menon P, Alderman H, Devakumar D, Fawzi W, Greenfield G, Hammoudeh W, He S, Lahiri A, Liu Z, Nguyen PH, Sethi V, Wang H, Neufeld LM, Patton GC. Strategies and interventions for healthy adolescent growth, nutrition, and development. Lancet. 2022 Jan 8;399(10320):198-210. doi: 10.1016/S0140-6736(21)01593-2. Epub 2021 Nov 29. PMID 34856192
- [Background] Hawkes C, Ruel MT, Salm L, Sinclair B, Branca F. Double-duty actions: seizing programme and policy opportunities to address malnutrition in all its forms. Lancet. 2020 Jan 11;395(10218):142-155. doi: 10.1016/S0140-6736(19)32506-1. Epub 2019 Dec 15. PMID 31852603
- [Background] Hawkes C, Demaio AR, Branca F. Double-duty actions for ending malnutrition within a decade. Lancet Glob Health. 2017 Aug;5(8):e745-e746. doi: 10.1016/S2214-109X(17)30204-8. Epub 2017 May 18. No abstract available. PMID 28528865
- [Background] WHO. Double-duty actions for nutrition. Policy Brief. Department of Nutrition for Health and Development World Health Organization. Geneva. Switzerland [Internet]. 2017. Available from: https://apps.who.int/iris/bitstream/handle/10665/255414/WHO-NMH-NHD-17.2-eng.pdf?ua=1 (Accessed on June 10, 2021)
- [Derived] Getacher L, Ademe BW, Belachew T. Effect of double duty interventions on dietary diversity score of adolescents using a cluster randomized controlled trial in Debre Berhan Regiopolitan City, Ethiopia. Sci Rep. 2025 Feb 13;15(1):5381. doi: 10.1038/s41598-025-88324-6. PMID 39948109
- [Derived] Getacher L, Ademe BW, Belachew T. Effect of double-duty interventions on double burden of malnutrition among adolescents in Debre Berhan Regiopolitan City, Ethiopia: a cluster randomised controlled trial. J Nutr Sci. 2024 Nov 28;13:e74. doi: 10.1017/jns.2024.68. eCollection 2024. PMID 39703895
- [Derived] Getacher L, Ademe BW, Belachew T. Double burden of malnutrition and its associated factors among adolescents in Debre Berhan Regiopolitan City, Ethiopia: a multinomial regression model analysis. Front Nutr. 2023 Jul 18;10:1187875. doi: 10.3389/fnut.2023.1187875. eCollection 2023. PMID 37545577